CLINICAL TRIAL: NCT00455858
Title: A 20-week, Multi-centre, Open-labelled, Non-comparative Evaluation of the Safety and Efficacy of Insulin Detemir in Combination With Oral Anti-diabetic Drug(s), in Subjects With Type 2 Diabetes Mellitus Who Were Inadequately Controlled on Current Therapy in Korea
Brief Title: Evaluation of the Glycaemic Control With Insulin Detemir as an add-on to Current Oral Anti-diabetic Drug Treatment in Subjects With Type 2 Diabetes in Korea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1762
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Results first posted 2010-02-23 (Estimated); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- insulin detemir (Active Comparator)
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Treat-to-target dose titration scheme, once daily, injected s.c. (under the skin).
  Other Names: Levemir®

SUMMARY:
This trial is conducted in Asia. This trial aims for evaluating the glycaemic control, measured as glycosylated haemoglobin (Hb1Ac), of once daily insulin detemir as an add-on to oral antidiabetic drug (OAD) in subjects with type 2 diabetes mellitus in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (diagnosed more than 12 months ago)
* HbA1c greater than 7.0 and less than 12.0% at screening
* Currently on any OAD in more than 3 months ago
* BMI (Body Mass Index) less than 35kg/m2

Exclusion Criteria:

* Previous treatment with insulin in more than 7 days within the last 3 months
* Uncontrolled treated/untreated hypertension (systolic blood pressure greater than 180mmHg and/or diastolic blood pressure less than 110mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Seoul, South Korea

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of eight study sites in South Korea.
Pre-assignment Details: Between screening and treatment with study drug, subjects were assessed for eligibility. After start of treatment, all subjects were to have their dosage titrated individually based on SMPG (self-monitored plasma glucose) values during the 20-week titration and treatment period to reach and maintain pre-breakfast SMPG below 6.0 mmol/L (108 mg/dL).
Groups:
- Insulin Detemir: Insulin detemir start dose of 0.2 U/kg body weight added to Subject's ongoing OAD (oral anti-diabetic drug) monotherapy or combination therapy of 2 or more OADs. Insulin detemir treatment is titrated based on subject's self-monitored plasma glucose.
Period: Overall Study
Arm/Group | Insulin Detemir
Started | 87 (Enrolled in study and exposed to study drug)
Completed | 81
Not Completed | 6
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 1
Not completed — Lack of Efficacy | 1
Not completed — Well controlled FPG without insulin | 1
Not completed — Withdrawal | 1

BASELINE CHARACTERISTICS:
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin A1c (HbA1c) at Week 20
Description: Change in Glycosylated Haemoglobin A1c (HbA1c) from baseline to week 20
Time Frame: week 0, week 20
Population: The analysis was based on Full Analysis Set (FAS) without any imputations. The definition of FAS is: All enrolled subjects exposed to at least one dose of study product and have at least one HbA1c data after 3 months being exposed to the study product.
Measure: Mean (Standard Deviation); unit: percentage change in HbA1c
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 81
percentage change in HbA1c
  HbA1c at baseline | 9.3 (1.1)
  HbA1c at week 20 | 8.2 (1.1)
  Change in HbA1c from baseline to week 20 | -1.2 (0.9)
Statistical Analysis 1: Comparison: Insulin Detemir; Test type: Superiority or Other; p < .0001, t-test; Least Square Mean = -1.356, 95% CI [-1.368 to -1.344]

2. Secondary Outcome: Change in Glycosylated Haemoglobin A1c (HbA1c) at Week 12
Description: Change in Glycosylated Haemoglobin A1c (HbA1c) at week 12 from baseline
Time Frame: week 0, week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change in HbA1c
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 82
percentage change in HbA1c
  HbA1c at baseline | 9.3 (1.1)
  HbA1c at week 12 | 8.2 (1.1)
  Change in HbA1c from baseline to week 12 | -1.2 (0.9)
Statistical Analysis 1: Comparison: Insulin Detemir; Test type: Superiority or Other; p < .0001, t-test; Least Square Mean = -1.338, 95% CI [-1.350 to -1.327]

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change in fasting plasma glucose (FPG) from baseline to week 12 and week 20
Time Frame: week 0, week 12, week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 85
mg/dL
  FPG at baseline, N=81 | 178 (54.2)
  FPG at week 12, N=77 | 118 (36.3)
  FPG at week 20, N=78 | 116 (35.8)
  Change in FPG from baseline to week 12, N=75 | -60 (55.8)
  Change in FPG from baseline to week 20, N=73 | -62 (61.5)
Statistical Analysis 1: Comparison: Insulin Detemir; Estimated mean decrease in FPG at week 12; Test type: Superiority or Other; p < .0001, Paired t-test; Least Square Mean = -69.553, 95% CI [-70.047 to -69.060]
Statistical Analysis 2: Comparison: Insulin Detemir; Estimated mean decrease in FPG at week 20; Test type: Superiority or Other; p < .0001, Paired t-test; Least Square Mean = -72.159, 95% CI [-72.647 to -71.671]

4. Secondary Outcome: Percentage of Subjects Achieving Glycosylated Haemoglobin A1c (HbA1c) Less Than 7.0%
Description: Percentage (%) of subjects achieving Glycosylated Haemoglobin A1c (HbA1c) treatment target levels less than 7.0%
Time Frame: week 12, week 20
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 85
percentage of participants
  Achieving HbA1c < 7% after 12 weeks, N=82 | 14.6
  Not achieving HbA1c < 7% after 12 weeks, N=82 | 85.4
  Achieving HbA1c < 7% after 20 weeks, N=81 | 12.3
  Not achieving HbA1c < 7% after 20 weeks, N=81 | 87.7

5. Secondary Outcome: Occurence of Hypoglycaemic Episodes
Description: Occurence of hypoglycaemic episodes - diurnal and nocturnal - over 20 weeks of treatment.
Time Frame: weeks 0-20
Population: For tabulating the occurence of hypoglycaemic episodes, the safety analysis set of all enrolled subjects exposed to at least one dose of study drug was used. For the adverse events, please refer to details in the adverse events section.
Measure: Number; unit: episodes
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 81
episodes
  Occurence of hypoglycaemic episodes: Diurnal | 92
  Occurence of hypoglycaemic episodes: Nocturnal | 78
  Occurence of hypoglycaemic episodes: Total | 170

ADVERSE EVENTS:
Time Frame: Adverse events were collected in a time span of 22 weeks.
Description: Safety analysis set contains all enrolled subjects exposed to at least one dose of study drug.
Arm/Group | Insulin Detemir
Serious Adverse Events (participants affected / at risk) | 5/87
Other Adverse Events (participants affected / at risk) | 15/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (N=87)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (N=87)
Nasopharyngitis (Infections and infestations) | 10 (10)
Upper respiratory tract infection (Infections and infestations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk acknowledges the Investigator's right to publish the entire results of the trial. Any such scientific paper, presentation, communication or other information concerning the investigation described in this protocol, should be submitted in writing to Novo Nordisk Trial Manager prior to submission for publication/presentation for comments. Comments will be given within four weeks from receipt of the manuscript.